CLINICAL TRIAL: NCT06611709
Title: Effectiveness of the Kinesiotaping in the Treatment of Chronic Lateral Epicondylitis: a Randomized, Sham-controlled, Single-blind Study
Brief Title: Effectiveness of the Kinesiotaping in the Treatment of Chronic Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ramazan Yılmaz, Associate Prof, Konya Beyhekim Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KonyaBeyhekimTRH2024
Record Dates: First submitted 2024-09-18; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Lateral Epicondylitis (tennis Elbow); Pain
Keywords: kinesiotaping; lateral epicondylitis; pain; exercises
MeSH Terms: conditions — Tennis Elbow; Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Kinesiotaping vs sham-taping
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kinesiotaping (Experimental): Kinesiotaping (real) + exercises
  Interventions: Device: Kinesiotaping: A standard 5-cm wide KinesioⓇ Tex Gold; Other: exercises
- Sham-taping (Sham Comparator): Sham-taping (non-elastic medical cloth tape) + exercises
  Interventions: Device: sham taping (non-elastic medical cloth tape); Other: exercises

INTERVENTIONS:
Device: sham taping (non-elastic medical cloth tape) — sham taping
  Arms: Sham-taping
Device: Kinesiotaping: A standard 5-cm wide KinesioⓇ Tex Gold — A standard 5-cm wide KinesioⓇ Tex Gold
  Arms: Kinesiotaping
Other: exercises — home-based exercises

SUMMARY:
Lateral epicondylitis significantly impacts daily activities and productivity at work, making it a condition of substantial clinical and socioeconomic importance.Despite its high prevalence, clinical significance, and impact on daily life, the optimal management of LE remains a topic of ongoing debate.

This study aims to investigate the efficacy of kinesiotaping (KT) on pain intensity, functional status, and quality of life in patients with chronic lateral epicondylitis (LE).

The study was conducted in the outpatient clinic for level 3 physical medicine and rehabilitation. Patients were randomized into two groups: the real kinesiotaping + home exercise group and the sham taping + home exercise group (randomized by a medical secretary outside the study). A set of widely accepted, literature-consistent primer and seconder outcomes were statistically compared to determine whether one treatment was superior to the other.

DETAILED DESCRIPTION:
Between February 1, 2024, and August 31, 2024, a total of 42 patients (17 females, 25 males) with chronic LE were included. Patients were randomized into either the KT or sham-controlled group. Patients were blinded to which group they were assigned to. The taping was performed by the same physician, who was trained and experienced in kinesiotaping.

Kinesiotaping and sham-taping were applied six times over three weeks. Both groups received recommendations for activity modification and a home-based stretching and strengthening exercise program. The exercise program was designed by an author who has a national book chapter on exercise for the treatment of lateral epicondylitis, taking into account patient specificity and adherence, and in accordance with the literaturExercise adherence was monitored through weekly outpatient controls (while taping) and by phone check-ins two weeks after the taping was completed.

Outcome measures were visual analog scale (VAS) pain score, Patient-Rated Forearm Evaluation Questionnaire (PRFEQ), grip strength, Disabilities of Arm, Shoulder, and Hand (DASH), quality of life in Short Form-36 (SF-36), and The Roles and Maudsley patient satisfaction score. The subjects were assessed before treatment, at the end of treatment (week three), and four weeks after the end of treatment (week seven).The assessment parameters were also conducted by the same researcher to ensure consistency.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* A pain severity of 4 or higher on the visual analog scale (VAS) during daily activities
* A history of lateral epicondylitis symptoms lasting at least three months

Exclusion Criteria:

* Communication difficulties
* Significant psychiatric disorders
* A history of trauma within the past six months
* Neuromuscular conditions
* Abnormalities of the upper limb
* Prior upper limb surgery
* A history of rheumatic diseases
* Cervical disc pathology, polyneuropathy, or hand disorders (such as carpal or cubital tunnel syndrome, de Quervain tenosynovitis, osteoarthritis)
* Receipt of any treatment for lateral epicondylitis (e.g., local injections, physical therapy, splints) within the last six month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Patient-Rated Tennis Elbow Evaluation Questionnaire (PRTEE) | baseline, week 3, and week 7
  0 (best) to 100 (worst)
VAS pain (0-10) | baseline, week 3, and week 7
  0 no pain; 10 unbearable/max. pain.

SECONDARY OUTCOMES:
The Disabilities of the Arm, Shoulder, and Hand (DASH) | baseline, week 3, and week 7
  0 (best condition) to 100 (worst condition)
grip strength | baseline, week 3, and week 7
  using a Jamar® dynamometer (in kilograms)
The Short Form-36 (SF-36) quality of life index | baseline, week 3, and week 7
  0, indicating the worst health status, to 100, representing the best possible health
Patient satisfaction/benefit scale (The Roles and Maudsley score) | baseline, week 3, and week 7
  The Roles and Maudsley score was utilized to evaluate pain and activity limitations in the assessment of treatment efficacy, categorized into four levels: 1 point indicating excellent, 2 points indicating good, 3 points indicating fair, and 4 points indicating poor.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Beyhekim Research and Training Hospital, Physical Medicine and Rehabilitation clinics, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Akkurt HE, Yilmaz R, Suna FS, Karpuz S, Yilmaz H. The effectiveness of kinesiotaping in treating chronic lateral epicondylitis: a randomized, sham-controlled, single-blind study. J Orthop Surg Res. 2025 Mar 14;20(1):274. doi: 10.1186/s13018-025-05658-7. PMID 40082899